CLINICAL TRIAL: NCT06258603
Title: The Effect of Oral Care Bundle Application on Salivary pH (Power of Hydrogen), Dry Mouth and Ventilator-associated Pneumonia in Intubated Patients
Brief Title: Oral Care of Intubated Intensive Care Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gül Güneş AKTAN, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-5T/40
Record Dates: First submitted 2023-12-19; First posted 2024-02-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia; Mechanical Ventilation Complication; Salivation; Dry Mouth
Keywords: oral health; oral care; intensive care; nursing; intubation; dry mouth
MeSH Terms: conditions — Pneumonia; Sialorrhea; Xerostomia | interventions — Patient Care Bundles

STUDY DESIGN:
Intervention Model Description: The randomization of the study was achieved by the faculty member of the University's Faculty of Medicine, Department of Biostatistics and Medical Informatics, with the R version 3.1.3 program. First of all, the individuals included in the study were stratified according to two age groups (19-44 years and 45-70 years) in the computer environment. Then, individuals in each age group were included in the experimental and control groups in a balanced manner using the block randomization method. The randomization list was hidden from the researcher and the patient and was given to the researcher by a third party during the application. Eligibility and randomization assessment was performed by a critical care nurse independent of the study.
Who Masked: Participant
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who received oral care bundle (Experimental): "A oral care bundle" protocol created by the researchers and it was applied by a researcher to experimental group.
  Interventions: Other: oral care bundle
- Patients receiving routine clinical oral care (Other): Routine oral care protocol used in intensive care unit was applied to control group by the patient's primary nurse.
  Interventions: Other: clinical oral care

INTERVENTIONS:
Other: oral care bundle — In the first stage, oral health was evaluated and data about the patient was collected.
  In the second stage, an oral care bundle containing an oral care combination was applied to the experimental group. According to this bundle application, patients were received tooth brushing (with chlorhexidine solution) and ice water application twice a day and moisturizing attempts 4 times a day.
  In the 3rd stage, saliva pH, dry mouth (amount of salivation) and ventilator associated pneumonia development status of the experimental group patients were evaluated.
  Measurements were made by the researcher using the Bedside Oral Exam scale, pH (power of hydrogen) strip and Schirmer Tear Test Strip.
  Data regarding whether patients were diagnosed with ventilator associated pneumonia were obtained from the Infection Control Committee.
  Arms: Patients who received oral care bundle
Other: clinical oral care — In the first stage, oral health was evaluated and data about the patient was collected.
  In the second stage, routine oral care protocol used in intensive care unit was applied to patients by the patients' primary nurse. According to this application, patients were received oral care using tongue depressor with wrapped in gauze and chlorhexidine solution 4 times a day.
  In the 3rd stage, saliva pH (power of hydrogen), dry mouth (amount of salivation) and ventilator associated pneumonia development status of the experimental group patients were evaluated.
  Measurements were made by the researcher using the Bedside Oral Exam scale, pH (power of hydrogen) strip and Schirmer Tear Test Strip.
  Data regarding whether patients were diagnosed with ventilator associated pneumonia were obtained from the Infection Control Committee.
  Arms: Patients receiving routine clinical oral care

SUMMARY:
The aim of the research was to examine the effect of oral care bundle application on oral health, salivary pH (power of hydrogen), dry mouth and ventilator associated pneumonia in intubated patients compared to standard oral care.

DETAILED DESCRIPTION:
Maintaining the integrity of the oral mucosa in intensive care unit patients is very important due to its close relationship with systemic health, disease risk and self-image, as well as comfort and nutrition. Serious problems develop in patients who have no or insufficient saliva movement or production, are unconscious, or have an artificial airway. Oral health problems, which begin with the deterioration of the saliva flow and content of intubated patients, lead to much more risky and costly situations that end in ventilator associated pneumonia. In the literature, it is seen that oral care practices performed in accordance with protocols increase the risk of complications and that bundle care practices used in different care areas increase the performance of care.In this randomized controlled study, people who were aged between 18 and 70, had received mechanical ventilation support, were intubated orally and in the first 24 hours of intubation, and had a stable hemodynamic status were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation support,
* orally intubation
* in the first 24 hours of intubation,
* stable hemodynamic status

Exclusion Criteria:

* pneumonia
* Sjögren's Syndrome,
* radiotherapy and/or chemotherapy,
* oral care contraindications,
* head and neck trauma,
* platelet count below 50 thousand,
* could not be positioned appropriately,
* agitation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Individual Identification Form | First day of data collection
  The form was prepared by the researcher in line with literature information. It consists of 9 questions covering the characteristics of the patients (demographic characteristics, diagnoses, APACHE II scores, Glasgow Coma Scale score, rules, feeding patterns, intubation tube number).
Bedside Oral Exam Scale | Evaluated for five days.
  Oral health was assessed using the scale. The scale consists of 8 subheadings (swallowing, lips, tongue, saliva, mucous membranes, gums, teeth or dentures, and smell). The scale score ranges from 8 points (perfect oral health) to 24 points (impaired oral health).
In this outcome measure, the patients'vsaliva pH (power of hydrogen) was evaluated. | The 1st, 3rd and 5th days of oral care practices
  Merck brand Universal pH 0-14 indicator was used to measure the saliva pH of the patients. The indicator was placed on the tongue and waited for 1 minute, and the resulting color change was compared with the color scale on the box. According to the literature, the average pH of unstimulated saliva has been determined to be approximately 6.8.
In this outcome measure, the patients' saliva amount was evaluated. | The 1st, 3rd and 5th days of oral care practices.
  Schirmer Tear Test Strip was used in the application. The Modified Schirmer Test strip was placed under the tongue by holding its end with forceps, and after waiting for 3 minutes, the mm value of the wetness on the strip was read.
In this outcome measure, it was evaluated whether ventilator-associated pneumonia occured in patients receiving care. | Evaluated for five days.
  To avoid bias regarding the method used, the diagnosis of ventilator associated pneumonia was made independently by the treatment team. In the Intensive Care Unit of Ege University Faculty of Medicine, Department of Anesthesiology and Reanimation, the diagnosis of ventilator associated pneumonia is made by the physician using the nosocomial infection diagnostic criteria of The Centers for Disease Control and Prevention (CDC). Information about the development of ventilator associated pneumonia was obtained from the infection control nurse.

CONTACTS AND LOCATIONS:
Locations (1):
- Gül Güneş AKTAN, Niğde, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Abdelhafez AI, Tolba AA. Nurses' practices and obstacles to oral care quality in intensive care units in Upper Egypt. Nurs Crit Care. 2023 May;28(3):411-418. doi: 10.1111/nicc.12736. Epub 2021 Dec 2. PMID 34855285
- [Background] Alja'afreh MA, Mosleh SM, Habashneh SS. The Effects of Oral Care Protocol on the Incidence of Ventilation-Associated Pneumonia in Selected Intensive Care Units in Jordan. Dimens Crit Care Nurs. 2019 Jan/Feb;38(1):5-12. doi: 10.1097/DCC.0000000000000334. PMID 30499786
- [Background] Andersson P, Persson L, Hallberg IR, Renvert S. Testing an oral assessment guide during chemotherapy treatment in a Swedish care setting: a pilot study. J Clin Nurs. 1999 Mar;8(2):150-8. doi: 10.1046/j.1365-2702.1999.00237.x. PMID 10401348
- [Background] Blot S, Deschepper M, Labeau S. De-adoption of chlorhexidine oral care and ICU mortality. Intensive Care Med. 2022 May;48(5):624-625. doi: 10.1007/s00134-022-06621-4. Epub 2022 Jan 17. No abstract available. PMID 35037992
- [Background] Chair SY, Chan DWK, Cao X. The interaction of subglottic drainage, cuff pressure, and oral care on endotracheal tube fluid leakage: A benchtop study. Aust Crit Care. 2020 Jul;33(4):358-363. doi: 10.1016/j.aucc.2019.05.002. Epub 2019 Jun 24. PMID 31248697
- [Background] Cuthbertson BH, Dale CM. Less daily oral hygiene is more in the ICU: yes. Intensive Care Med. 2021 Mar;47(3):328-330. doi: 10.1007/s00134-020-06261-6. Epub 2020 Oct 10. No abstract available. PMID 33037882
- [Background] Dale CM, Rose L, Carbone S, Pinto R, Smith OM, Burry L, Fan E, Amaral ACK, McCredie VA, Scales DC, Cuthbertson BH. Effect of oral chlorhexidine de-adoption and implementation of an oral care bundle on mortality for mechanically ventilated patients in the intensive care unit (CHORAL): a multi-center stepped wedge cluster-randomized controlled trial. Intensive Care Med. 2021 Nov;47(11):1295-1302. doi: 10.1007/s00134-021-06475-2. Epub 2021 Oct 5. PMID 34609548